CLINICAL TRIAL: NCT02085460
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase 2 Trial of Rebamipide Liquid to Determine the Effective Dose for Prevention of Chemoradiotherapy-induced Oral Mucositis in Patients With Head and Neck Cancer
Brief Title: A Phase 2 Trial of Rebamipide Liquid to Determine the Effective Dose for Prevention of Chemoradiotherapy-induced Oral Mucositis in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 037-12-001; JapicCTI-142467 (Other: Japic)
Record Dates: First submitted 2014-03-11; First posted 2014-03-12 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): 6 times daily
  Interventions: Drug: Placebo
- 2% Rebamipide liquid (Experimental): 6 times daily
  Interventions: Drug: 2% Rebamipide liquid
- 4% Rebamipide liquid (Experimental): 6 times daily
  Interventions: Drug: 4% Rebamipide liquid

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: 2% Rebamipide liquid
  Arms: 2% Rebamipide liquid
Drug: 4% Rebamipide liquid
  Arms: 4% Rebamipide liquid

SUMMARY:
To investigate the efficacy and safety of rebamipide liquid for chemoradiotherapy-induced oral mucositis in patients with head and neck cancer following administration of rebamipide and to determine the optimal dose of rebamipide.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients scheduled for definitive or postoperative chemoradiotherapy.
* Patients with a histopathological diagnosis of head and neck cancer and primary tumor in one of the following regions.

  1. Definitive therapy: nasopharynx, oropharynx, hypopharynx, or larynx
  2. Postoperative therapy: oral cavity, oropharynx, hypopharynx, or larynx
* Patients with no history of chemotherapy, radiotherapy, or chemoradiotherapy for head and neck cancer
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Patients who are able to hold fluid in the mouth
* Patients who are able to swallow the investigational medicinal product (IMP)
* Patients expected to survive for at least 3 months
* Patients who have given written informed consent in person
* Patients who can stay at or visit the hospital for scheduled examinations and observations
* Patients who are able to take contraceptive measures to avoid pregnancy of the patient or their partner from the time of informed consent until 4 weeks after completion of IMP administration

Exclusion Criteria:

* Patients with primary malignant tumors other than head and neck cancer.
* Patients with symptomatic viral, bacterial, or fungal infection
* Patients with serious renal impairment
* Patients with distant metastasis
* Patients with severe complications (uncontrolled cardiac disease, diabetes, hypertension, etc)
* Patients with any of the following laboratory test results:

  1. Neutrophil count: <1500 L
  2. Platelet count: <75000 L
  3. Hemoglobin: <10.0 g/L
  4. Aspartate aminotransferase (AST): >3 times the upper limit of the reference value at the trial site
  5. Alanine aminotransferase (ALT): >3 times the upper limit of the reference value at the trial site
  6. Serum bilirubin: >1.5 times the upper limit of the reference value at the trial site
  7. Serum albumin: <3.0 g/dL
  8. Serum creatinine: >1.5 the upper limit of the reference value at the trial site
  9. Creatinine clearance : <30 mL/min
* Patients complicated with autoimmune disease
* Patients requiring continuous systemic administration of glucocorticoid
* Female patients who are pregnant or lactating, who may possibly be pregnant, or who wish to become pregnant
* Patients who have participated in any other clinical trial within 4 weeks prior to initiation of chemoradiotherapy
* Patients who have a history of drug allergy to rebamipide, cisplatin, or other platinum compounds
* Patients who are otherwise judged by the investigator or sub-investigator to be inappropriate for inclusion in the trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-ichi Hashimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (5):
- Japan (5):
  - Chubu Region
  - Chugoku Region
  - Kanto Region
  - Kinki Region
  - Tohoku Region

REFERENCES:
- [Background] Ueno T, Zenda S, Konishi T, Yurikusa T, Shibasaki Y, Nagamoto H, Fujii M. The post hoc analysis comparing the severity grades of chemoradiotherapy-induced oral mucositis scored between the central and local assessors in a multicenter, randomized controlled trial of rebamipide for head and neck cancer. Int J Clin Oncol. 2019 Mar;24(3):241-247. doi: 10.1007/s10147-018-1355-7. Epub 2018 Nov 13. PMID 30426268
- [Derived] Yokota T, Ogawa T, Takahashi S, Okami K, Fujii T, Tanaka K, Iwae S, Ota I, Ueda T, Monden N, Matsuura K, Kojima H, Ueda S, Sasaki K, Fujimoto Y, Hasegawa Y, Beppu T, Nishimori H, Hirano S, Naka Y, Matsushima Y, Fujii M, Tahara M. Efficacy and safety of rebamipide liquid for chemoradiotherapy-induced oral mucositis in patients with head and neck cancer: a multicenter, randomized, double-blind, placebo-controlled, parallel-group phase II study. BMC Cancer. 2017 May 5;17(1):314. doi: 10.1186/s12885-017-3295-4. PMID 28476132

RESULTS

PARTICIPANT FLOW:
Groups:
- 2% Rebamipide Liquid; 4% Rebamipide Liquid; Placebo: 6 times daily (The treatment started 3 days prior to the initiation of chemoradiotherapy and continued for another 77 days.)
Period: Overall Study
Arm/Group | 2% Rebamipide Liquid | 4% Rebamipide Liquid | Placebo
Started | 31 | 32 | 31
Completed | 17 | 24 | 21
Not Completed | 14 | 8 | 10
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Physician Decision | 1 | 1 | 2
Not completed — Withdrawal by Subject | 11 | 5 | 7

BASELINE CHARACTERISTICS:
Population: Full analysis set comprised patients who received the study drug or placebo at least once and whose efficacy data were collected immediately after beginning the treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2% Rebamipide Liquid | 4% Rebamipide Liquid | Placebo | Total
Number analyzed (Participants) | 31 | 32 | 31 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 19 | 55
  >=65 years | 14 | 13 | 12 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 17
  Male | 26 | 26 | 25 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 31 | 32 | 31 | 94
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 31 | 32 | 31 | 94

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade ≥3 Oral Mucositis Determined by Clinical Examination and Assessed by Central Review According to the Common Terminology Criteria of Adverse Events (CTCAE) Version 3.0.
Description: Investigators who had undergone specific training assessed the severity of oral mucositis twice every week. To evaluate the severity of oral mucositis objectively, the clinical findings of the oral mucosa as well as functional disorders and symptomatic aspects were recorded in the Oral Mucositis Assessment Sheet by each investigator. Photographic documentation of the oral mucosa was also submitted by each investigator, 3 days before or 57 days after initiation of chemoradiotherapy, or at the time of withdrawal. The Oral Mucositis Assessment Sheets and photographic documentation were then reviewed by the Oral Mucositis Evaluation Committee to grade the severity of oral mucositis according to the CTCAE 3.0.z
Time Frame: 77 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | 2% Rebamipide Liquid | 4% Rebamipide Liquid | Placebo
Number analyzed (Participants) | 31 | 32 | 31
percentage of participants | 29.0 | 25.0 | 38.7

2. Secondary Outcome: Number of Subjects Who Did Not Developed Grade ≥3 Mucositis
Description: Day 1 was defined as the start of chemotherapy.
Time Frame: Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 77
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | 2% Rebamipide Liquid | 4% Rebamipide Liquid | Placebo
Number analyzed (Participants) | 31 | 32 | 31
participants
  Day 1 | 31 | 31 | 31
  Day 8 | 29 | 31 | 30
  Day 15 | 27 | 30 | 29
  Day 22 | 25 | 29 | 23
  Day 29 | 23 | 25 | 23
  Day 36 | 20 | 20 | 19
  Day 43 | 18 | 18 | 16
  Day 50 | 17 | 18 | 15
  Day 57 | 12 | 16 | 13
  Day 64 | 11 | 15 | 11
  Day 71 | 8 | 13 | 8
  Day 77 | 6 | 11 | 8

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from start of the study drug administration up to Day 85
Description: Safety set comprised those who received the study drug or placebo at least once and whose safety data were collected at least once after beginning the treatment.
Arm/Group | 2% Rebamipide Liquid | 4% Rebamipide Liquid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 5/31 | 5/32 | 4/31
Other Adverse Events (participants affected / at risk) | 31/31 | 32/32 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2% Rebamipide Liquid (N=31) | 4% Rebamipide Liquid (N=32) | Placebo (N=31)
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Pharyngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2% Rebamipide Liquid (N=31) | 4% Rebamipide Liquid (N=32) | Placebo (N=31)
Anaemia (Blood and lymphatic system disorders) | 7 | 9 | 10
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 2 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 27 | 30 | 30
Nausea (Gastrointestinal disorders) | 25 | 24 | 25
Constipation (Gastrointestinal disorders) | 21 | 25 | 24
Dry mouth (Gastrointestinal disorders) | 20 | 24 | 19
Vomiting (Gastrointestinal disorders) | 9 | 13 | 12
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 10
Dysphagia (Gastrointestinal disorders) | 4 | 5 | 6
Cheilitis (Gastrointestinal disorders) | 3 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 2 | 0 | 0
Malaise (General disorders) | 14 | 12 | 14
Fatigue (General disorders) | 0 | 6 | 4
Oedema peripheral (General disorders) | 2 | 5 | 3
Pyrexia (General disorders) | 1 | 4 | 2
Face oedema (General disorders) | 2 | 2 | 0
Infusion site extravasation (General disorders) | 0 | 3 | 1
Thirst (General disorders) | 0 | 0 | 2
Vessel puncture site inflammation (General disorders) | 2 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1 | 1
Hypersensitivity (General disorders) | 1 | 2 | 0
Oral candidiasis (Infections and infestations) | 6 | 12 | 7
Pharyngitis (Infections and infestations) | 4 | 3 | 4
Device related infection (Infections and infestations) | 0 | 1 | 2
Influenza (Infections and infestations) | 1 | 0 | 2
Rhinitis (Infections and infestations) | 2 | 0 | 1
Lung infection (Infections and infestations) | 2 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 2 | 0
Staphylococcal infection (Infections and infestations) | 0 | 2 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 22 | 26 | 20
Wound complication (Injury, poisoning and procedural complications) | 1 | 2 | 1
Weight decreased (Investigations) | 15 | 12 | 18
White blood cell count decreased (Investigations) | 12 | 12 | 12
Neutrophil count decreased (Investigations) | 9 | 8 | 9
Lymphocyte count decreased (Investigations) | 9 | 9 | 6
Blood creatinine increased (Investigations) | 5 | 4 | 3
Platelet count decreased (Investigations) | 3 | 4 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0
Weight increased (Investigations) | 2 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 0
C-reactive protein increased (Investigations) | 1 | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 21 | 22 | 23
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 4 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 5 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 4 | 3 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 4 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 22 | 26 | 25
Headache (Nervous system disorders) | 1 | 1 | 4
Somnolence (Nervous system disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 6 | 6 | 4
Renal impairment (Renal and urinary disorders) | 5 | 5 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 11 | 15 | 10
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 7 | 7
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No